CLINICAL TRIAL: NCT06684236
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Sleeping After General Anesthesia in Elderly Patients Undergoing Abdominal Surgery
Brief Title: Acupoint Stimulation and Postoperative Sleep in Elderly Patients
Acronym: ASIS-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XJH-A-20240627
Record Dates: First submitted 2024-07-05; First posted 2024-11-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Sleep
Keywords: acupoint stimulation; general anesthesia; sleep; elderly patients
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint stimulation (Experimental): transcutaneous electrical acupoint stimulation is one of the many forms of acupuncture, and is a distinctive part of Chinese medicine that has been practiced in China for thousands of years. It is employed by placing electrodes on acupoint and electrical stimulation is given after anesthetic induction to the end of the surgery
  Interventions: Other: transcutaneous electrical stimulation; Other: electrodes attachment
- Control (Sham Comparator): Electrodes are placed on same acupoints as the experimental group, and will receive the "optimal intensity test" before the anesthesia induction, but no electrical stimulation is given during the operation
  Interventions: Other: electrodes attachment

INTERVENTIONS:
Other: transcutaneous electrical stimulation — electrical stimulation is given through electrodes attached to the skin
  Arms: Acupoint stimulation
Other: electrodes attachment — electrodes are attached to the skin area of Neiguan acupoint, which is located on 3cm above the transverse crease of the wrist

SUMMARY:
Sleeping model can be affected after surgery. Anesthetics may be involved in the change. The changing of sleeping mode may exert adverse effect on postoperative recovery. Acupuncture and related techniques has been used for treating sleeping disorder. In this study, the effect of transcutaneous electrical acupoint stimulation on sleeping model after general anesthesia will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Age≥65 years old
* scheduled for abdominal surgery under general anesthesia

Exclusion Criteria:

* anticipated duration of surgery longer than 5 hours or shorter than 1 hour
* American society of anesthesiologists status over stage 3
* Participants with sleep apnea or moderate and severe obstructive sleep apnea syndrome (defined by Apnea Hypopnea Index (AHI))
* Participants with preoperative sleep disturbances (diagnostic criteria of sleep disturbances according to the International Classification of Sleep Disorders, Third Edition (ICSD-3))
* Participants with a history of alcohol or drug abuse
* Participants with severe hepatic or renal insufficiency kidney disease
* Participants with contraindications to the use of acupoint stimulation (including those with infection or injury of the skin to attach electrodes, and those with implanted electronic devices)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
total sleeping time during the first postoperative night | the first postoperative night, on an average of 12 hours

SECONDARY OUTCOMES:
Total sleep time during the first 24 hours after surgery | from discharge from post-anesthesia care unit to 24 hours later, totally 24 hours
The Epworth Sleepiness Scale (ESS) score at 24 hours after surgery | 24 hours after surgery
The Athens Insomnia Scale (AIS) score at 24 hours after surgery | 24 hours after surgery
The Athens Insomnia Scale (AIS) score at 48 hours after surgery | 48 hours after surgery
The Epworth Sleepiness Scale (ESS) score at 48 hours after surgery | 48 hours after surgery
The Athens Insomnia Scale (AIS) score at discharge from hospital | the last day before discharge from hospital, at an average of 12 hours
The Epworth Sleepiness Scale (ESS) score at discharge from hospital | the last day before discharge from hospital, at an average of 12 hours
sleep efficiency(%) during the first postoperative night | the first postoperative night, at an average of 12 hours
  sleep efficiency is defined as the ratio of total sleep time to time in bed
duration of rapid eye movement sleep during the first postoperative night | the first postoperative night, at an average of 12 hours
  The unit of duration of rapid eye movement sleep is by minutes
number of wake during the first postoperative night | the first postoperative night, at an average of 12 hours
incidence of delirium during hospitalization | From end of surgery to discharge from hospital, assessed up to 7 days
length of postoperative hospital stay | From end of surgery to discharge from hospital, at an average of 5 days
number of needs for rescue analgesia by 24 hours after surgery | from discharge from operation room to 24 hours later, totally 24 hours
Number of participants with major complications during hospitalization, including cardiac failure, cardiac infarction, respiratory failure | From end of surgery to discharge from hospital, assessed up to 7 days
Scale of quality of recovery at discharge from hospital | the last day before discharge from hospital, at an average of 12 hours
  Scale of quality of recovery is measured by the Quality-of-recovery 15 item scale (QoR-15)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu WT, Hsu CM, Hung SC, Hung SY. Acupuncture Improves Sleep Disorders and Depression among Patients with Parkinson's Disease: A Meta-Analysis. Healthcare (Basel). 2023 Jul 17;11(14):2042. doi: 10.3390/healthcare11142042. PMID 37510483
- [Background] El Iskandarani S, Sun L, Li SQ, Pereira G, Giralt S, Deng G. Acupuncture improves certain aspects of sleep in hematopoietic stem cell transplantation patients: a secondary analysis of a randomized controlled trial. Acupunct Med. 2023 Dec;41(6):319-326. doi: 10.1177/09645284231181403. Epub 2023 Jul 6. PMID 37409464